CLINICAL TRIAL: NCT06799299
Title: Diagnostic Performance of the Inferior Vena Cava Collapsibility to Predict Fluid Responsiveness in Early Post-kidney Transplantation Period
Brief Title: Collapsibility Index of the Inferior Vena Cava and Kidney Transplantation
Acronym: CIVC-KT
Status: Not yet recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PS25002
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Fluid Responsiveness in Early Post-kidney Transplantation Period
Keywords: Inferior vena cava; Fluid responsiveness; Fluid overload; Delayed graft function; Kidney transplantation
MeSH Terms: conditions — Edema; Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: cardiac output increases by >10%.
  Interventions: Other: No Intervention
- Non-responders: cardiac output increases by ≤10%.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
Delayed graft function following renal transplantation is common occurrence and is associated with an increased risk of acute rejection and chronic allograft nephropathy. Post transplant patients are usually hyperhydrated to optimize renal blood flow and thus graft function. However, cardiac failure to respond adequately to volume expansion can lead to renal venous congestion and visceral interstitial sodium and water overload, both of which are associated with the delayed kidney graft function. To our knowledge, no predictive index for fluid responsiveness has been evaluated in post-renal transplantation setting. In intensive care, the inferior vena cava variability index measured by transthoracic echocardiography (TTE) under standardized breathing conditions, is a simple, non-invasive and effective tool for predicting fluid responsiveness in patients hospitalized for sepsis. Applying this index in the post-renal transplantation period could potentially optimize early management and enhance the recovery of kidney graft function.

In this study, we aim to evaluate the diagnostic performance of the inferior vena cava variability index in predicting fluid responsiveness after renal transplantation. This is a monocentric, prospective, and observational study conducted in the nephrology intensive care unit at University Reims Hospital.

DETAILED DESCRIPTION:
The study is a prospective, observational, single-center cohort (nephrology intensive care unit at University Reims Hospital) designed to evaluate the diagnostic performance of the Inferior Vena Cava Variability Index (IVCv) in predicting fluid responsiveness in post-kidney transplantation patients.

The study aims to decrease the number of patients delayed graft function and to optimize recovery of kidney function. Delayed graft function is a frequent complication occurring in 20-25% of kidney transplants. Delayed graft function increases the risk of acute rejection and chronic graft dysfunction. Fluid management is critical in the early postoperative period to optimize renal blood flow and graft function, but excessive fluid administration in non-responsive patients can lead to renal congestion and interstitial edema, negatively impacting graft recovery.

The IVCv, a simple and non-invasive echocardiographic index, assesses the diameter variability of the inferior vena cava induced by respiratory pressure changes. This index has been validated in septic patients to predict fluid responsiveness following volume expansion but has not yet been evaluated in the specific context of kidney transplantation. This study hypothesizes that IVCv could predict fluid responsiveness in this population, enabling tailored fluid management.

The primary objective of this study is therefore to determine the diagnostic performance of the inferior vena cava variability to predict fluid responsiveness in early post-kidney transplantation period.

Secondary objectives include:

1. Evaluating the diagnostic performance of central venous pressure variability (CVPv) to predict fluid responsiveness in early post-kidney transplantation period.
2. Identifying predictive markers of non-responsiveness to volume expansion.
3. Assessing renal response to fluid responsiveness.
4. Investigating associations between non-responsiveness, delayed graft function, and intra-abdominal pressure variations.

Key procedures involve transthoracic echocardiography (TTE) before and after fluid administration. Parameters such as IVCv, cardiac output, and central venous pressure will be systematically measured. Additional monitoring includes daily renal function markers, urine output, and extracellular hydration status during the first month post-transplantation.

The study will enroll 150 adult end-stage renal disease patients undergoing kidney transplantation at CHU Reims. Fluid responsiveness is defined as a ≥10% increase in cardiac output following a 500 mL crystalloid infusion. Non-responders are patients with <10% cardiac output improvement.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of End-stage renal disease (ESRD)
* Hospitalization in the nephrology intensive care unit at Reims University Hospital
* Hospitalization due to renal transplantation
* Willingness to provide informed consent and participate in the study
* Receiving volume expansion following renal transplantation.

Exclusion criteria:

* Inability to obtain high-quality ultrasound images
* Unavailability of Intra-vesical pressure and central venous pressure measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered to all eligible patients during the preoperative phase of renal transplantation in the nephrology intensive care unit of REIMS hospital. Eligibility will be confirmed based on clinical, biological and immunological assessments demonstrating the feasibility of the transplant. Patients will receive detailed information about the study's objectives and procedures through an information leaflet. Those who agree to participate will be included in the study.
  Each patient's participation will extend from Day 0 of the transplant procedure to Month 1post transplant.
  All patients requiring a post transplantation volume expansion will be included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Inferior vena cava variability index (IVCv) and the cardiac output (to determine diagnostic performances of this index) | Day 1
  IVCv will be measured by echocardiography before the volume expansion Patients will be classified as responders if their cardiac output increases by > 10% after volume expansion, and in non-responders if not

SECONDARY OUTCOMES:
Central venous pressure variability index and the cardiac output (to determine diagnostic performances of this index) | Day 1
  Central venous pressure variability index before the volume expansion
Predictive markers of non-responsiveness to volume expansion | Day 1
  Patients' characteristics at baseline and the cardiac output
Renal response to fluid responsiveness | Day 30
  Changes in plasma creatinine levels, diuresis and intra-abdominal pressure after volume expansion
Intra-abdominal pressure variations | Day 30
  Associations between non-responsiveness, delayed graft function, and intra-abdominal pressure variations

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France